CLINICAL TRIAL: NCT04057300
Title: Ticagrelor Compared to Clopidogrel in Acute Coronary Syndromes - the TC4 Comparative Effectiveness Study
Brief Title: Ticagrelor Compared to Clopidogrel in Acute Coronary Syndromes
Acronym: TC4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, James Brophy, Principle Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TC4/2019-4530
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Acute Coronary Syndrome
Keywords: Cardiovascular disease; Myocardial Infarction; Stroke; Clopidogrel; Ticagrelor; Platelet Aggregation Inhibitors; Pragmatic Trial
MeSH Terms: conditions — Acute Coronary Syndrome; Cardiovascular Diseases; Myocardial Infarction; Stroke | interventions — Ticagrelor; Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ticagrelor 90mg (Experimental): Ticagrelor: 180 mg loading dose followed by 90 mg BID. Aspirin: 325 loading dose followed by 81 mg daily.
  Interventions: Drug: Ticagrelor 90mg; Drug: acetylsalicylic acid (ASA) 81mg
- Clopidogrel 75mg (Active Comparator): Clopidogrel: 300 mg loading dose followed by 75 mg daily. Aspirin: 325 loading dose followed by 81 mg daily.
  Interventions: Drug: Clopidogrel 75mg; Drug: acetylsalicylic acid (ASA) 81mg

INTERVENTIONS:
Drug: Ticagrelor 90mg — Ticagrelor tablet
  Other Names: Brilinta
  Arms: Ticagrelor 90mg
Drug: Clopidogrel 75mg — Clopidogrel tablet
  Other Names: Plavix
  Arms: Clopidogrel 75mg
Drug: acetylsalicylic acid (ASA) 81mg — acetylsalicylic acid tablet
  Other Names: Aspirin

SUMMARY:
The McGill University Health Center (MUHC) Division of Cardiology, with funding from the Canadian Institute of Health Research, is performing this randomized controlled trial to determine which dual antiplatelet therapy (DAPT), ticagrelor + aspirin (T+A) or clopidogrel and aspirin (C+A), is the most effective and safest for our patients. While the PLATO trial reported that T+A was superior, the prespecified group of North American patients (about 1/10 of the total study sample) actually did better with C+A, although this difference was not statistically significant. When the FDA approved T, they also stated: "Lack of Robustness of PLATO Superiority with Failure in the US Makes a Confirmatory Study Mandatory." As no confirmatory study has been done, this TC4 study aims to fill that void.

Study design: A cluster randomization design, so all patients will receive either T+A or C+A, depending on the month they arrive at the MUHC when they start their DAPT. We will follow patients through their electronic health records. The patients have no follow-up visits for this research project.

DETAILED DESCRIPTION:
Acute Coronary Syndrome (ACS) is most often caused by erosion or rupture of an atherosclerotic plaque associated with inflammation, thrombus formation, vasoconstriction, and microembolisation. In unremitting circumstances, thrombosis at the site of plaque rupture or erosion leads to complete compromise of coronary blood flow and ultimately myocardial infarction (MI). Platelet adhesion, activation and aggregation, therefore, play key roles in the transformation of a stable atherosclerotic plaque to an unstable lesion and antiplatelet drugs have become a mainstay in the prevention of recurrent cardiovascular events.

A large multicenter RCT (PLATO) showed a statistically significant decrease in composite CV outcomes with the newer ticagrelor compared to clopidogrel. This has prompted both European and Canadian guideline writers to endorse ticagrelor/aspirin as the DAPT of choice. However residual uncertainties regarding the choice of DAPT are highlighted by the PLATO subgroup analysis that showed an increased risk with ticagrelor in North America (NA) patients. This led to delayed FDA approval, dissenting FDA reviews and a reluctance in US guidelines to recommend the ticagrelor DAPT regime over others.

The main area of uncertainty, at least from the NA perspective, hinges on the small number of NA patients randomized in the PLATO trial and their increased risk with ticagrelor (n=1814, HR 1.25; 95% CI 0.93 - 1.67). The risk in NA patients was statistically significantly different from the benefit seen in the other subgroups (P=0.04) and the crux of the debate is then whether to believe the subgroup analysis or the combined study results (n=18624, HR, 0.84; 95% CI 0.77 to 0.92). The complete study provides maximal information but perhaps at a cost of being less representative of what to expect in NA practice. Conventional statistical paradigms would say that given the pre-specified nature of the geographic subgroup analysis and given the statistically significant interaction observed, one should concentrate on the subgroup results and not the combined results.

The conventional statistical model used in the PLATO analysis subsumes that every patient, regardless of differences in recruitment characteristics or ancillary treatment strategies received in the different regions, is completely identical in their response to the studied intervention. It seems highly unlikely that patients from the 43 PLATO enrolling countries are truly identical in their drug response given recruitment, genetic and background treatment variations.

This project will resolve these uncertainties and address the crucial clinical question of which DAPT regime is best after an ACS? This proposal will double the currently available evidence with a novel research design using inexpensive, electronic data and will provide a feasible answer to this important clinical question.

More information can be found here:

https://brophyj.github.io/index.html

ELIGIBILITY:
Inclusion Criteria:

* Patients that are prescribed a dual-antiplatelet therapy (DAPT) regimen following an acute coronary syndrome (ACS) event.
* ACS, with or without ST-segment elevation.
* STEMI and NSTEMI positive biomarkers and appropriate ECG changes will be required.
* NSTEMI patients with negative biomarkers are generally considered as unstable angina and will also be eligible for study inclusion if their treating physician has determined that DAPT is appropriate.
* Patients provided written informed consent.

Exclusion Criteria:

* A decision from the patients attending physician to circumvent randomization and assign the patient a specific dual-antiplatelet therapy regimen.
* A contraindication to clopidogrel or ticagrelor
* Patients diagnosed with chronic total occlusion percutaneous coronary intervention (CTO PCI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1038 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
The hazard ratio for the number of participants that develop the outcome, a composite of cardiovascular-related mortality, myocardial infarction (MI), or stroke. | 12 months
  ICD-10 Codes

SECONDARY OUTCOMES:
The primary outcome (The hazard ratio for the number of participants that develop the outcome, a composite of cardiovascular-related mortality, myocardial infarction (MI), or stroke) stratified by sex. | 12 months
The hazard ratio for the number of participants that develop the outcome, a composite of cardiovascular-related mortality, myocardial infarction (MI), or stroke. | 36 months
The primary outcome (The hazard ratio for the number of participants that develop the outcome, a composite of cardiovascular-related mortality, myocardial infarction (MI), or stroke) stratified by sex | 36 months
The hazard ratio for the number of participants with any cardiovascular-related mortality event | 12 months
The hazard ratio for the number of participants with any acute MI event | 12 months
The hazard ratio for the number of participants with any stroke event | 12 months
The hazard ratio for the number of participants with any major bleeding requiring hospitalization event | 12 months
The hazard ratio for the number of participants with any recurrent coronary revascularization(s) event | 12 months
The hazard ratio for the number of participants with any reported drug side effects | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: James Brophy, MD, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valgimigli M, Bueno H, Byrne RA, Collet JP, Costa F, Jeppsson A, Juni P, Kastrati A, Kolh P, Mauri L, Montalescot G, Neumann FJ, Petricevic M, Roffi M, Steg PG, Windecker S, Zamorano JL, Levine GN; ESC Scientific Document Group; ESC Committee for Practice Guidelines (CPG); ESC National Cardiac Societies. 2017 ESC focused update on dual antiplatelet therapy in coronary artery disease developed in collaboration with EACTS: The Task Force for dual antiplatelet therapy in coronary artery disease of the European Society of Cardiology (ESC) and of the European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2018 Jan 14;39(3):213-260. doi: 10.1093/eurheartj/ehx419. No abstract available. PMID 28886622
- [Background] Mehta SR, Bainey KR, Cantor WJ, Lordkipanidze M, Marquis-Gravel G, Robinson SD, Sibbald M, So DY, Wong GC, Abunassar JG, Ackman ML, Bell AD, Cartier R, Douketis JD, Lawler PR, McMurtry MS, Udell JA, van Diepen S, Verma S, Mancini GBJ, Cairns JA, Tanguay JF; members of the Secondary Panel. 2018 Canadian Cardiovascular Society/Canadian Association of Interventional Cardiology Focused Update of the Guidelines for the Use of Antiplatelet Therapy. Can J Cardiol. 2018 Mar;34(3):214-233. doi: 10.1016/j.cjca.2017.12.012. Epub 2017 Dec 19. PMID 29475527
- [Background] Levine GN, Bates ER, Bittl JA, Brindis RG, Fihn SD, Fleisher LA, Granger CB, Lange RA, Mack MJ, Mauri L, Mehran R, Mukherjee D, Newby LK, O'Gara PT, Sabatine MS, Smith PK, Smith SC Jr. 2016 ACC/AHA Guideline Focused Update on Duration of Dual Antiplatelet Therapy in Patients With Coronary Artery Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2016 Sep 6;68(10):1082-115. doi: 10.1016/j.jacc.2016.03.513. Epub 2016 Mar 29. No abstract available. PMID 27036918
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Background] Center for Drug Evaluation and Research. Complete Response Review Addendum Sponsor Safety Reporting Submissions: NDA 22-433 and IND 65,808 SD 632 Drug: ticagrelor (BrilintaTM). 2011. https://wwwaccessdatafdagov/drugsatfda_docs/nda/2011/022433Orig1s000MedRpdf.
- [Derived] Kutcher SA, Dendukuri N, Dandona S, Nadeau L, Brophy JM. Ticagrelor Compared to Clopidogrel in Acute Coronary Syndromes trial (TC4): a Bayesian pragmatic cluster randomized controlled trial. CMAJ. 2025 Mar 30;197(12):E309-E318. doi: 10.1503/cmaj.241862. PMID 40164463